CLINICAL TRIAL: NCT03904927
Title: Role of Local Therapy for Patients with Oligorecurrent and Oligometastatic Esophageal Squamous Cell Carcinoma After Radical Treatment: a Prospective, Randomized Phase II Clinical Study
Brief Title: Local Therapy for Oligorecurrent and Oligometastatic Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai13
Record Dates: First submitted 2019-03-28; First posted 2019-04-05 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Oligorecurrent and Oligometastatic Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Radiation; Surgical Procedures, Operative; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): The arm will be treated with combined systemic therapy and local therapy such as radiation, surgery or radiofrequency ablation.
  Interventions: Other: Radiation, Surgery or Radiofrequency ablation; Drug: Systemic therapy
- Control Arm (Active Comparator): The arm will be treated with systemic therapy alone.
  Interventions: Drug: Systemic therapy

INTERVENTIONS:
Other: Radiation, Surgery or Radiofrequency ablation — Patients with no more than 4 metastases located in less than 3 organs/ lymphatic drainage regions treated with combined systemic therapy and radiation, surgery or radiofrequency.
  Arms: Experimental Arm
Drug: Systemic therapy — 1. First-line chemotherapy (previously without chemotherapy), paclitaxel 175mg/m2, d1+cisplatin 25mg/m2, d1-3, repeated every 28 days, intravenous infusion, a total of 4 cycles.
  2. If patients have a history of chemotherapy, use a regimen of docetaxel 75mg/m2, d1, intravenous infusion, repeated every 21 days for a total of 4 cycles. If previously use docetaxel but not irinotecan, then use a regimen of irinotecan 180mg/m2, d1, d15, repeated every 28 days for a total of 4 cycles. If both docetaxel and irinotecan have been used, the investigator could decide the chemotherapy regimen.
  3. Anti-PD1 antibodies plus chemotherapy could be used as first-line systemic therapy and Anti-PD1 antibodies could be used as second-line therapy.

SUMMARY:
The aim of the study is to determine if intervening with combined local therapy and chemotherapy prior to chemotherapy alone in patients with oligorecurrent and oligometastatic esophageal squamous cell carcinoma led to significant improvements in progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with oligometastatic diseases and pathologically confirmed esophageal squamous cell carcinoma after initial radical treatment [i.e., completely resected surgery or radical (chemo)radiotherapy], the primary esophageal sites are controlled.

   Note:
   1. Definition of metastasis: patients with distant organ metastases or non-regional lymph node metastases; or patients with distant organs/non-regional lymph node metastases and regional lymph node metastases as defined in the eighth edition of the AJCC. Patients with only regional lymph node metastasis and/or anastomotic/esophageal recurrence are not eligible for enrollment.
   2. According to the classification of oligometastatic disease, oligometastasis including synchronous oligometastasis, metachronous oligometastasis, and repeat oligometastasis could be enrolled in this trial.
   3. In visceral metastases or non-regional lymph node metastases, at least one metastatic lesion obtains pathological confirmation.
2. The total number of metastases is 4 or less and maximum 3 metastases in any single organ system (i.e. lung, liver). The maximum diameter for each lesion should be no more than 5 cm.

   1. Each lesion was counted separately at the time of registration and contributed to the total number of metastases.If regional recurrences are existed, all positive regional lymph nodes are count together as one lesion. For non-regional lymph node metastases, adjacent metastatic lymph nodes can be treated as one lesion.
   2. Lesions that have subsided during previous treatment (i.e., were no longer visible on CT or had eliminated affinity on PET-CT) are not included in the total number. For patients with synchronous oligometastasis, the controlled primary tumor and regional lymph nodes on imaging are counted toward the total of 4.
3. All metastases of current diagnosis did not receive local treatment such as radiotherapy, surgery, radiofrequency ablation before enrollment.
4. Previous chemotherapy was allowed, but no anti-tumor medication was received within 3 months prior to the start of treatment.
5. The measurable lesion was determined by the investigator based on the RECIST 1.1 assessment. A lesion located in a previous radiotherapy area can be considered a target lesion if it is confirmed to progress and is considered to be measurable according to RECIST 1.1.
6. The patient is over 18 years old and has an ECOG score of 0-1.
7. Estimated survival time >12 weeks.
8. The function of vital organs meets the following requirements:

   1. Neutrophil absolute count (ANC) ≥ 1.5 × 10^9 / L
   2. platelets ≥ 100 × 10^9 / L;
   3. Hemoglobin ≥ 9g / dL;
   4. serum albumin ≥ 2.8g / dL;
   5. Total bilirubin ≤ 1.5 × ULN, ALT, AST and / or AKP ≤ 2.5 × ULN; if there is liver metastasis, ALT and / or AST ≤ 5 × ULN; if there is liver metastasis or bone metastasis AKP ≤ 5 × ULN;
   6. serum creatinine ≤ 1.5 × ULN or creatinine clearance > 60 mL / min;
   7. For patients with pulmonary lesions or previous lung irradiation who are known or suspected to have impaired lung function, the forced expiratory volume (FEV1) for 1 second of lung function must be above 1L.
9. Female subjects of childbearing age must have a negative urine or serum pregnancy test within 72 hours prior to randomization. Subjects agreed to adequate contraception during the trial.
10. The patient is voluntarily enrolled and obtained the informed consent form signed by the patient or his legal representative.

Exclusion Criteria:

1. Primary tumor of esophagus is confirmed uncontrolled or progressive by imaging or gastroscope,or any esophageal or nodal recurrence locates in the previous radiation field.
2. The pathological diagnosis of any metastatic lesion is clearly different from the primary tumor or diagnosed as a second primary tumor.
3. Patients participated in any investigational drug study within 4 weeks preceding the start of treatment.
4. If there is a metastasis within 3 months after definitive treatment, or the number of metastases is more than 4.
5. Patients with uncontrolled brain metastases, or vertebral body metastasis with spinal cord compression symptoms.
6. The toxicity of previous anti-tumor treatment has not recovered to ≤ National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 level 1 (except for hair loss) or the level specified by the inclusion/exclusion criteria.
7. Patients with uncontrolled pleural, pericardial or pelvic effusion that requires repeated drainage.
8. Patients who have received chemotherapy, anti-tumor medication, major surgery or severe trauma within 3 months before enrollment.
9. Pregnant or breastfeeding women.
10. Patients with history of immunodeficiency, or severe medical diseases that are not well controlled, which may have effect on the treatment of this study.
11. Any other malignant tumor was diagnosed within 5 years prior to or after the diagnosis of ESCC, except for malignant tumors with a low risk of metastasis and death (5-year survival rate >90%), such as well-treated basal cells or squamous cell skin cancer or cervical cancer in situ.
12. The investigator judged that patients could not cooperate with the treatment, or have other factors that might cause him to be forced to terminate the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Time from the date of randomisation to the date of progression or date of death from any cause, whichever came first, assessed up to 3 years
  progression-free survival will be measured as time to either progression or death

SECONDARY OUTCOMES:
Overall survival | The survival time from the date of randomisation to the date of death from any cause, assessed up to 3 years
  Overall survival will be measured as time to death from any cause.
Local control | the time from the date of randomisation to the date of local failure or the last follow-up, assessed up to 3 years
  Local control will be measured as time to local recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Universtiy Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Q, Chen J, Lin Y, Ye J, Shen W, Luo H, Li B, Huang W, Wei S, Song J, Wang Y, Yang H, Lai S, Zhu H, Ai D, Chen Y, Deng J, Hao S, Zhao K. Systemic therapy with or without local intervention for oligometastatic oesophageal squamous cell carcinoma (ESO-Shanghai 13): an open-label, randomised, phase 2 trial. Lancet Gastroenterol Hepatol. 2024 Jan;9(1):45-55. doi: 10.1016/S2468-1253(23)00316-3. Epub 2023 Nov 18. PMID 37980921
- [Derived] Liu Q, Chen J, Li B, Ye J, Wei S, Wang Y, Yang H, Zhu Z, Lai S, Li L, Chen Y, Wang J, Xiang J, Zhao K. Local therapy for oligometastatic esophageal squamous cell carcinoma: a prospective, randomized, Phase II clinical trial. Future Oncol. 2021 Apr;17(11):1285-1293. doi: 10.2217/fon-2020-0873. Epub 2021 Feb 25. PMID 33626929